CLINICAL TRIAL: NCT05341635
Title: Innovative Method for the Rapid and Low-cost Search of SARS-CoV-2 in Respiratory Samples: Validation With Multiple Diagnostic Systems and Process Automation.
Brief Title: FAst and SimplE COVID-19 Causing Virus SARS-CoV-2 Detection
Acronym: FASE2
Status: Completed | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Collaborators: Azienda Ospedaliera San Gerardo di Monza (Other); University of Milan (Other); A.O. Ospedale Papa Giovanni XXIII (Other)
Responsible Party: Sponsor
Other Study IDs: FASE2
Record Dates: First submitted 2021-04-21; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; Molecular; Diagnostic; Test
MeSH Terms: conditions — COVID-19; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal and saliva specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 Symptomatic inpatients: Patients admitted to the Unit of Infectious Diseases of the ASST Monza for COVID-19 will run the collection of a nasopharyngeal swab, performed as part of the normal diagnostic routine; will take up to two samples collected in parallel to the development and optimization of the new method/process preanalitico and for the clinical validation of the performance of the pre-analytic method. The subjects will be adequately informed, both verbally and by means of a summary document of the study before signing a consent for participation in the study.
  Interventions: Diagnostic Test: Swab sampling
- COVID-19 Suspected subjects: To the subjects who present at the Emergency department of the ASST Monza for symptomatology referable to the COVID-19 and to patients on discharge from the Unit of Infectious Diseases of the ASST Monza for complete healing from COVID-19 will run the collection of a nasopharyngeal swab, performed as part of the normal diagnostic routine; will take up to two samples collected in parallel to the development and optimization of the new method/process preanalitico and for the clinical validation of the performance of the pre-analytic method. The subjects will be adequately informed, both verbally and by means of a summary document of the study before signing a consent for participation in the study.
  Interventions: Diagnostic Test: Swab sampling

INTERVENTIONS:
Diagnostic Test: Swab sampling — Collection of three nose-pharyngeal and oral swabs

SUMMARY:
Observational study using biological material. The group of subjects in the study is represented by 100 male and female patients hospitalized with COVID-19 symptomatology and 100 non-hospitalized subjects with suspected COVID-19 diagnosis for a total of 200 patients.

The expected recruitment time is about 6 months.

DETAILED DESCRIPTION:
Clinical study using biological material. The group of subjects in the study is represented by 100 male and female patients hospitalized with COVID-19 symptomatology and 100 non-hospitalized subjects with suspected COVID-19 diagnosis for a total of 200 patients.

The expected recruitment time is about 6 months. Each patient will be carried out a nasopharyngeal swab in UTM medium™ which will be tested according to the diagnostic procedure in use, a second nasopharyngeal swab resuspended in MSwab™ and a third oral dry swab that will be transported to the laboratory of Clinical Microbiology and Virology of UNIMIB and resuspersed in the MSwab™ transport medium. The samples will then be treated according to the new workflow defined by the pilot study, i.e. optimization of alternative sample transport systems, in combination with a rapid method of viral RNA extraction, and evaluation of viral inactivation at the end of the extraction phase, by viral culture at the BSL3 laboratory of the Virology laboratory of the University of Milan.

The samples collected and transported on UTM™ medium will be sent to the Microbiology Laboratory of the ASST of Monza and analyzed through the NIMBUS-Seegene platform as per diagnostic routine.

The residual volume of the UTM™ medium sample and all remaining samples taken by each patient will be sent to the Laboratory of Microbiology and Clinical Virology of the University of Milano-Bicocca to be processed through the new preanalytic method in combination with different analytical kits.

A percentage of each sample will be sent to the Virology Laboratory of the University of Milan for testing using the analytical protocol suggested by the CDC.

The study samples will also be used for the validation of a new innovative analytical test for SARS-CoV-2, in Real-Time Multiplex One- Step PCR, developed to be combined with the preanalytic process with thermal extraction, fast and low cost, with high-throughput automation.

All residual volumes of the samples in the study, and related nucleic acids, will be rated and stored in Bio-Bank according to international "standard operating procedures" the validation of further and/or new diagnostic tests for the search for for SARS-CoV-2 (ASST PG23 in collaboration with BBMRI.it).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the U.O. of Infectious Diseases of the San Gerardo Hospital in Monza with documented COVID-19 symptomatology;
* COVID-19 asymptomatic or post-hospital discharge;
* People of legal age;
* Patients who agree to participate have given their consent by signing a specially prepared form.

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The group of study subjects is represented by 100 men and women patients hospitalized with COVID-19 symptoms and 100 non-hospitalized subjects with suspected COVID-19 diagnosis for a total of 200 patients.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Development of a rapid, safe and simplified diagnostic method for the molecular detection and quantification of SARS-CoV-2 in respiratory samples through the set-up of a Real-Time PCR assay expressing results in viral genomic copies/microL of sample | Up to three months
  Comparison between the preanalytical procedures commonly used for the processing of the nasopharyngeal swab in the search for SARS-CoV-2 and faster, lower cost and less expensive procedures for the material used as reagents and consumables
Clinical validation of the performance of the preanalytic method (medium selection and nucleic acids extraction method) in combination with analytical Real-Time PCR assay | Through study completation, an average of 6 months
  Clinical validation of new preanalytical and detection processes, in comparison with different commercial kits in use in Lombardy region laboratories
Development and validation of new preanalytic and analytical methods integrated with high-throughput automation. | Through study completation, an average of 6 months
  Optimization of all the preanalytical and analytical aspects of a diagnostic path for the search of SARS-CoV-2 from different swabs and scale-up of executable samples per day through the implementation of high-throughput processing instrumentation.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera San Gerardo Monza, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: Undecided